CLINICAL TRIAL: NCT00305136
Title: Advancement of Psychophysics of Pain Modulation From Lab to Clinic: Constructing Susceptibility Profile for Appearance of Postoperative Neuropathic Pain
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Israel Scientific Foundation (Unknown)
Responsible Party: Principal Investigator, d_yarnitsky, Head of Neurology department, Rambam Health Care Campus
Other Study IDs: Thoracotomy02CTIL; ISF
Record Dates: First submitted 2006-03-19; First posted 2006-03-21 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Pain, Postoperative
Keywords: thoracotomy; post-operative pain; chronic pain; endogenous analgesia; temporal summation; central sensitization; prediction; Patients Who Should Undergo Thoracotomy
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recent advances in the field of pain psychophysics that have enhanced the understanding of pain processing by the nervous system seem to characterize the individual pattern of pain processing, thereby enabling the prediction of a person's susceptibility to develop chronic pain consequent to surgery.

In this project, the researchers propose to apply a wide array of advanced testing methods in order to prospectively assess the pain modulation pattern of pain free patients about to undergo an elective thoracotomy. Since about half of post-thoracotomy patients suffer from chronic neuropathic postoperative pain, the researchers expect to identify which tests predict a risk for this pain and the relative power of the relevant tests in this prediction, and to construct a short and applicable tool, the 'pain susceptibility profile', that will reliably predict the risk for the development of pain. The expected results of this project will serve the field of pain prevention by identifying patients at risk and tailoring interventions to reduce the risk of chronic pain.

DETAILED DESCRIPTION:
The common prevalence of painful syndromes following surgical interventions and injuries calls for a preventive therapeutic approach that can only be based on better insight into the pain modulation mechanisms in these patients. Recent advances in the field of pain psychophysics that have enhanced our understanding of pain processing by the nervous system seem to characterize the individual pattern of pain processing, thereby enabling the prediction of a person's susceptibility to develop chronic pain consequent to surgery.

In this project, we propose to apply a wide array of advanced testing methods in order to prospectively assess the pain modulation pattern of pain free patients about to undergo an elective thoracotomy. Tests will include:

1. psychophysical tests: pain thresholds and suprathreshold magnitude estimation, temporal summation, endogenous analgesia - diffuse noxious inhibitory control (DNIC);
2. tests for the interaction between pain and the autonomic nervous system including the inhibitory effect of vagal activation on pain perception, and the response pattern of the sympatho-parasympathetic balance to noxious stimulation; and
3. evaluation of personality components known to be associated with chronic pain including anxiety, catastrophization and somatization.

Since about half of post-thoracotomy patients suffer from chronic neuropathic postoperative pain, we expect to identify which tests predict a risk for this pain and the relative power of the relevant tests in this prediction, and to construct a short and applicable tool, the 'pain susceptibility profile', that will reliably predict the risk for the development of pain. The contribution of the above tests to the severity of acute postoperative pain, and of the latter on the development of the chronic postoperative pain will also be evaluated.

The expected results of this project will serve pain prevention by identifying patients at risk and tailoring interventions to reduce the risk of chronic pain. Also, in the wider pain research context, this understanding will allow better design and analysis of studies on pain mechanisms and therapies by considering the pain susceptibility of participating patients.

ELIGIBILITY:
Inclusion Criteria:

* Pain free patients to undergo major thoracic operation with both malignant and non-malignant diseases.

Exclusion Criteria:

* Psychiatric or cognitive dysfunction precluding use of psychophysics
* Existing thoracic pain
* Patients who cannot communicate in Hebrew

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Pain free patients to undergo major thoracic operation with both malignant and non-malignant diseases.
  Exclusion Criteria:
  * Psychiatric or cognitive dysfunction precluding use of psychophysics
  * Existing thoracic pain
  * Patients who cannot communicate in Hebrew
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Yarnitsky, Professor, Principal Investigator — Neurology Department Chairman, Rambam Medical Center, Haifa, Israel
Locations (1):
- Rambam Medical Center, Haifa, Israel